CLINICAL TRIAL: NCT00340184
Title: A Phase II Trial of Radiation Therapy With Concurrent Paclitaxel/Carboplatin Chemotherapy in High-risk Cervical Cancer Patients After Radical Hysterectomy
Brief Title: A Safety and Efficacy of CCRT With Paclitaxel/Carboplatin as Adjuvant Therapy to Post-operative Cervical Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Korean Gynecologic Oncology Group (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KGOG1001
Record Dates: First submitted 2006-06-20; First posted 2006-06-21 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2006-01

CONDITIONS: Cervical Cancer
Keywords: concurrent; chemoradiation; paclitaxel; carboplatin
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — CP protocol

INTERVENTIONS:
Drug: paclitaxel, carboplatin

SUMMARY:
The purpose of this study is to determine whether post-operative concurrent chemoradiation with paclitaxel/carboplatin is effective and safe in the treatment of high risk cervical cancer patients.

DETAILED DESCRIPTION:
Stage Ib to IIa cervical cancer can be treated effectively with either radioterapy or radical hysterectomy plus pelvic lymph node dissection. However, several pathological risk factors have been identified to compromise the treatment outcome. They include lymph node metastasis, the involvement of vaginal resection margin, and the parametrial invasion. In these patients, postoperative RT is commonly recommended and has been demonstrated to improve the local control, but not survival rate. Recently, It is reported that the additon of concurrent chemotherapy to postoperative RT reduced pelvic failures and enhanced progression free survival. In addition, paclitaxel/platinum combination chemotherapy was demonstrated to have superior progression-free survical over single agent platinum in a primary treatment of stage IV or recurrent cervical cancer.

Based on this obseration, we evaluated the efficacy and safety of CCRT with paclitaxel/carboplatin in patients with postoperative high risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients undertaken radical hysterectomy with diagnosis of invasive cervical cancer Ib-IIa (non-small cell type)
* Patients must have at least one of the following risk factors; pelvic lymph node involvemet, involvement of vaginal resection margin,parametrial invasion.
* Patients must have a GOG performance of 0, 1, or 2.
* Patients must have expected life span over 6 months.

Exclusion Criteria:

* Patients with peripheral neurotoxicity over grade 2 in CTC criteria.
* Patients with history of chemotherapy or radiation treatment.
* Patients with histologicallly proven or highly suspected metastasis to paraaortic lymph node.
* Patients with history of hypersensitive reaction to platinum agent.

Ages: 20 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Enrollment: 55
Dates: Start 2004-08

PRIMARY OUTCOMES:
Two year disease free survival

SECONDARY OUTCOMES:
5 year overall survical, toxicity profile

CONTACTS AND LOCATIONS:
Overall Officials: Soon Beom Kang, Professor, Study Chair — Korean Gynecologic Oncology Group
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee TS, Kang SB, Kim YT, Park BJ, Kim YM, Lee JM, Kim SM, Kim YT, Kim JH, Kim KT. Chemoradiation with paclitaxel and carboplatin in high-risk cervical cancer patients after radical hysterectomy: a Korean Gynecologic Oncology Group study. Int J Radiat Oncol Biol Phys. 2013 Jun 1;86(2):304-10. doi: 10.1016/j.ijrobp.2013.01.035. PMID 23642625